CLINICAL TRIAL: NCT05007730
Title: Enhancing Health and Quality of Life for Individuals With Dementia Through Transitional-State Snacks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Collaborators: Oregon Health and Science University (Other); Oregon Partnership for Alzheimer's Research (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02042020.009
Record Dates: First submitted 2021-07-28; First posted 2021-08-16 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Dementia; Nutrition Poor
Keywords: Caregiver
MeSH Terms: conditions — Dementia; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental)
  Interventions: Dietary Supplement: Transitional-state food therapeutic nutrition supplement

INTERVENTIONS:
Dietary Supplement: Transitional-state food therapeutic nutrition supplement — Participants will consume at least one "snack-sized" package of the transitional-state food supplements per day across the intervention trial.

SUMMARY:
Malnutrition significantly contributes to the disability and mortality associated with Alzheimer's disease and Alzheimer's disease-related dementias. Thus, nutritional status is one important, modifiable clinical factor for maintaining physical and cognitive health among persons with dementia (PWD). This project will pilot an innovative approach to enhancing nutrition through the use of transitional-state snack supplements, or foods that start as one texture and change to another.

Specifically, this study aims to demonstrate the feasibility, acceptability, and safety of a transitional-state therapeutic nutrition supplement among adults with dementia. The central hypothesis is that access to ready-made, savory, nutrient- dense snack supplements that resemble "typical" preferred foods and eating habits will result in improved nutritional intake and status among PWD.

ELIGIBILITY:
Inclusion Criteria:

* Medically stable
* Community dwelling
* Has a medical diagnosis of dementia or possible dementia

Exclusion Criteria:

* Does not live at home
* Cannot participate in the protocol independently and do not have a consistent caregiver who can provide assistance
* Does not have smartphone access
* Requires 100% feeding assistance
* Is NPO (nil per os)
* Has multiple food allergies
* Requires a strict renal, low-fat, and/or no-salt diet
* Is deemed unsafe for the transitional-state foods by a speech-language pathologist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-11-03 (Actual); Study Completion 2025-11-03 (Actual)

PRIMARY OUTCOMES:
Participant enrollment rates (%) | Measured during recruitment (at baseline, prior to study onset; week 0)
  The percentage of participants enrolled (i.e., who meet all eligibility criteria) as compared to the total number of participants who are recruited (i.e., initiate contact with the research team)
Proportion of participants deemed eligible to consume transitional-state foods | Prior to enrollment (to determine eligibility at baseline, prior to study onset; week 0)
  Instrumental swallowing assessments will be conducted for each participant by a licensed speech-language pathologist to determine whether the potential participant can safely consume transitional-state foods based on their swallowing physiology. The number of potential participants deemed eligible to consume this consistency of food will be compared to the total number of potential participants receiving the swallow study.
Participant retention rates (%) | Measured at the end of the study (post-intervention, after 8 weeks of snack consumption)
  The percentage of participants retained (i.e., who who remain enrolled and participate for the duration of the study) as compared to the total number of participants who are enrolled
Change in acceptability of nutrition supplements | Measured weekly for enrolled participants (weeks 1, 2, 3, 4, 5, 6, 7, 8)
  Using a Likert (5 point) rating scale, participants will rate their acceptability of the nutrition supplements each week. Change in acceptability will be calculated over the length of the study (e.g., increased or decreased acceptability over time)
Number of test snacks consumed each week | Measured weekly for enrolled participants (weeks 1, 2, 3, 4, 5, 6, 7, 8)
  As a measured of adherence to the protocol, participants will document the total number of test snacks consumed each week (protocol is for at least one snack per day)

SECONDARY OUTCOMES:
Change in malnutrition status (not present, present, moderate, severe) | Measured at baseline (study onset) and post-intervention (end of study after 8 weeks of snack consumption)
  Malnutrition status (not present, present, moderate, severe) will be assessed via a nutrition-focused physical exam (NFPE) by a registered dietitian. The exams will be guided by the recommendations of the American Society for Parenteral and Enteral Nutrition (ASPEN) in conjunction with the Academy of Nutrition and Dietetics (AND) and use the following characteristics for diagnosing malnutrition: insufficient energy intake, weight loss, loss of muscle mass, loss of subcutaneous fat, fluid accumulation, and diminished functional status. Using published definitions of the six clinical characteristics, a diagnosis of severe malnutrition, moderate malnutrition, or not malnourished will be made.
Change in malnutrition risk score | Measured at baseline (study onset) and post-intervention (end of study after 8 weeks of snack consumption)
  A malnutrition risk score will be calculated using the Mini Nutritional Assessment-Short Form (MNA-SF). Using the information collected by a registered dietitian during a nutrition-focused physical exam, the MNA-SF will be scored; the MNA-SF is a six-item, validated, and reliable screening tool for malnutrition risk.
Change in daily energy intake (kcal/d) | Baseline (study onset), mid-intervention (approximately 4 weeks into the trial), post-intervention (end of study after 8 weeks of snack consumption)
  Daily energy intake (in kcal/d) will be calculated based on photo-assisted, 24-hour dietary recalls completed via telephone. Three recalls will take place over the course of 2 weeks for each time point of interest.
Change in fat intake (g/d) | Baseline (study onset), mid-intervention (approximately 4 weeks into the trial), post-intervention (end of study after 8 weeks of snack consumption)
  Daily fat intake (in g/d) will be calculated based on photo-assisted, 24-hour dietary recalls completed via telephone. Three recalls will take place over the course of 2 weeks for each time point of interest.
Change in protein intake (g/d) | Baseline (study onset), mid-intervention (approximately 4 weeks into the trial), post-intervention (end of study after 8 weeks of snack consumption)
  Daily protein intake (in g/d) will be calculated based on photo-assisted, 24-hour dietary recalls completed via telephone. Three recalls will take place over the course of 2 weeks for each time point of interest.
Change in carbohydrate intake (g/d) | Baseline (study onset), mid-intervention (approximately 4 weeks into the trial), post-intervention (end of study after 8 weeks of snack consumption)
  Daily carbohydrate intake (in g/d) will be calculated based on photo-assisted, 24-hour dietary recalls completed via telephone. Three recalls will take place over the course of 2 weeks for each time point of interest.
Change in calcium intake (mg/d) | Baseline (study onset), mid-intervention (approximately 4 weeks into the trial), post-intervention (end of study after 8 weeks of snack consumption)
  Daily calcium intake (in mg/d) will be calculated based on photo-assisted, 24-hour dietary recalls completed via telephone. Three recalls will take place over the course of 2 weeks for each time point of interest.
Change in vitamin D intake (mg/d) | Baseline (study onset), mid-intervention (approximately 4 weeks into the trial), post-intervention (end of study after 8 weeks of snack consumption)
  Daily vitamin D intake (in mg/d) will be calculated based on photo-assisted, 24-hour dietary recalls completed via telephone. Three recalls will take place over the course of 2 weeks for each time point of interest.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Oregon, Eugene, Oregon
  - Oregon Health & Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barewal R, Shune S, Ball J, Kosty D. A Comparison of Behavior of Transitional-State Foods Under Varying Oral Conditions. Dysphagia. 2021 Apr;36(2):316-324. doi: 10.1007/s00455-020-10135-w. Epub 2020 May 26. PMID 32458146